CLINICAL TRIAL: NCT01185509
Title: A Phase II, Single Arm, Open Label Study to Evaluate the Efficacy and Safety of Trastuzumab and Vinorelbine in Advanced Breast Cancer Patients With Human Epidermal Growth Factor-2 (HER2) Negative Primary Tumors and HER2 Positive Circulating Tumor Cells
Brief Title: Trastuzumab and Vinorelbine in Advanced Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Not enough confirmed responses to continue treatment.
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Beth Israel Deaconess Medical Center (Other); Massachusetts General Hospital (Other); Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Ian E. Krop, MD, PhD, Assistant Professor of Medicine, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-207; H4913s (Other: Genentech, Inc)
Record Dates: First submitted 2010-08-18; First posted 2010-08-20 (Estimated); Results first posted 2017-05-24 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Breast Cancer; Metastatic Breast Cancer
Keywords: HER2 negative; HER2 positive
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Vinorelbine

STUDY DESIGN:
Intervention Model Description: The analysis was performed for 2 separate cohorts due to a change in study conduct during the trial (see arm description).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Trastuzumab and Vinorelbine - Cohort A (Experimental): Cycle 1: Patients received trastuzumab 8 mg/kg intravenously (IV) on day 1 and vinorelbine 25 mg/kg IV on days 1, 8 and 15 of each 21 day cycle Cycles 2+: Patients received trastuzumab 6 mg/kg IV on day 1 and vinorelbine 25 mg/kg IV on days 1, 8 and 15 of each 21 day cycle Patients were treated until disease progression or unacceptable toxicity. Eligibility required patients to have HER2 amplification by fluorescence in situ hybridization (FISH) (mean ratio > 2.0). The CTC tests of the first 11 patients were done at DFCI. The study team then decided to proceed with a different CTC test performed outside of DFCI. Because the method of CTC isolation was different from that performed by DFCI, the first 11 patients were placed into a separate cohort (Cohort A) and the remaining 20 patients represented the main cohort.
  Interventions: Drug: trastuzumab; Drug: vinorelbine
- Trastuzumab and Vinorelbine - Main Cohort (Experimental): Cycle 1: Patients received trastuzumab 8 mg/kg intravenously (IV) on day 1 and vinorelbine 25 mg/kg IV on days 1, 8 and 15 of each 21 day cycle Cycles 2+: Patients received trastuzumab 6 mg/kg IV on day 1 and vinorelbine 25 mg/kg IV on days 1, 8 and 15 of each 21 day cycle Patients were treated until disease progression or unacceptable toxicity. Eligibility required patients to have HER2 amplification by FISH (mean ratio > 2.0). The CTC tests of the first 11 patients were done at DFCI. The study team then decided to proceed with a different CTC test performed outside of DFCI. Because the method of CTC isolation was different from that performed by DFCI, the first 11 patients were placed into a separate cohort (Cohort A) and the remaining 20 patients represented the main cohort.
  Interventions: Drug: trastuzumab; Drug: vinorelbine

INTERVENTIONS:
Drug: trastuzumab
Drug: vinorelbine
  Other Names: navelbine

SUMMARY:
The purpose of this research study is to see what effects trastuzumab in combination with vinorelbine has on breast cancer when the participant has circulating tumor cells that are positive for the protein called HER2. Trastuzumab is an FDA approved drug that targets HER2. The drug combination of trastuzumab and vinorelbine is an effective treatment for patients with breast cancers that are positive for HER2. This trial seeks to determine if the combination can also benefit participants whose original breast cancer was HER2 negative but whose circulating tumor cells are HER2 positive.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the objective response rate (ORR) of trastuzumab and vinorelbine in patients with metastatic breast cancer with HER2 negative primary tumors and HER2 positive circulating tumor cells.

Secondary

* To describe the number of CTCs and the CTCs characteristics before and after therapy, and to explore the correlation of these findings with response.
* To further characterize the safety and tolerability.
* To evaluate progression-free survival.
* To evaluate clinical benefit rate [complete response (CR)+partial response (PR)+stable disease (SD)>24 weeks].

Exploratory

* To determine the clinical feasibility of high-throughput mutation profiling on circulating tumor cells (CTCs).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic invasive mammary carcinoma. The primary cancer must be HER2 negative by fluorescence in situ hybridization and/or immunohistochemistry.
* Patients must have CTCs with HER2 amplification by FISH.
* Measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension as 20mm or greater with conventional techniques of as 10mm or greater with spiral CT scan.
* Study participants must have either archival primary tumor or metastatic tumor tissue available to allow analysis to confirm their HER2 status.
* Patients must have received at least 1 prior chemotherapy regimen for metastatic breast cancer or evidence of disease progression within 6 months of completing adjuvant chemotherapy. Patients can receive any number of biological or hormonal regimens and remain eligible.
* 18 years of age or older
* Life expectancy of greater than 3 months
* ECOG Performance Status of 0, 1 or 2
* Normal organ and marrow function as outlined in the protocol
* Women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation.

Exclusion Criteria:

* Participants must have recovered from all reversible toxicities related to prior therapy before beginning protocol treatment, and may not have any pre-existing treatment-related toxicities in excess of grade 2
* Participants may not be receiving any other investigational agents while participating in this study
* Participants may not have received trastuzumab or vinorelbine in the past
* Participants receiving any medications or substances that are inhibitors of cytochrome P450 isoenzymes in the CYP3A subfamily are ineligible.
* EKG abnormalities of known clinical significance, such as prolonged QT.
* Left ventricular ejection fraction < 50%
* Patients with peripheral neuropathy of any etiology that exceeds grade 1 are ineligible
* Uncontrolled intercurrent illness
* Individuals with symptomatic or progressive brain metastases are ineligible. Subjects with treated brain metastases are eligible if they have no radiographic or other signs of progression in the brain for 1 month or longer after completion of local therapy. Any corticosteroid use for brain metastases must have been discontinued without subsequent appearance of symptoms for more than 4 weeks prior to study treatment.
* Individuals with active second malignancy are ineligible. Patients that are disease-free from a previously treated non-breast malignancy and have a 20% or less chance of recurrence are eligible.
* Pregnant or breast feeding women
* HIV-positive individuals on combination antiretroviral therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian Krop, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Parsons HA, Macrae ER, Guo H, Li T, Barry WT, Tayob N, Wulf GM, Isakoff SJ, Krop IE. Phase II Single-Arm Study to Assess Trastuzumab and Vinorelbine in Advanced Breast Cancer Patients With HER2-Negative Tumors and HER2-Positive Circulating Tumor Cells. JCO Precis Oncol. 2021 Nov;5:896-903. doi: 10.1200/PO.20.00461. PMID 34994617

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients enrolled from November 2010 through July 2014.
Groups:
- Trastuzumab and Vinorelbine - Cohort A; Trastuzumab and Vinorelbine - Main Cohort: Cycle 1: Patients received trastuzumab 8 mg/kg intravenously (IV) on day 1 and vinorelbine 25 mg/kg IV on days 1, 8 and 15 of each 21 day cycle Cycles 2+: Patients received trastuzumab 6 mg/kg IV on day 1 and vinorelbine 25 mg/kg IV on days 1, 8 and 15 of each 21 day cycle Patients were treated until disease progression or unacceptable toxicity. Eligibility required patients to have HER2 amplification by FISH (mean ratio > 2.0). The CTC tests of the first 11 patients were done at DFCI. The study team then decided to proceed with a different CTC test performed outside of DFCI. Because the method of CTC isolation was different from that performed by DFCI, the first 11 patients were placed into a separate cohort (Cohort A) and the remaining 20 patients represented the main cohort.
Period: Overall Study
Arm/Group | Trastuzumab and Vinorelbine - Cohort A | Trastuzumab and Vinorelbine - Main Cohort
Started | 11 | 20
Completed | 0 (Since treatment was not of fixed duration, all participants were considered as 'Not Completed'.) | 0 (Since treatment was not of fixed duration, all participants were considered as 'Not Completed'.)
Not Completed | 11 | 20
Not completed — Progression/Relapse | 9 | 15
Not completed — Physician Decision | 2 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Death | 0 | 1
Not completed — Intercurrent Illness | 0 | 1

BASELINE CHARACTERISTICS:
Population: The analysis dataset is comprised of all treated patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Trastuzumab and Vinorelbine - Cohort A | Trastuzumab and Vinorelbine - Main Cohort | Total
Number analyzed (Participants) | 11 | 20 | 31
Age, Continuous [Median (Full Range); unit: years] | 50 [26 to 78] | 54 [34 to 66] | 54 [26 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 20 | 31
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 20 | 31
Estrogen Receptor Status at Metastatic Diagnosis [Count of Participants; unit: Participants]
  Positive | 9 | 8 | 17
  Negative | 2 | 5 | 7
  Unknown | 0 | 7 | 7
Progesterone Receptor Status at Metastatic Diagnosis [Number; unit: participants]
  Positive | 4 | 4 | 8
  Negative | 7 | 9 | 16
  Unknown | 0 | 7 | 7

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of patients achieving complete response (CR) or partial response (PR) based on RECIST 1.1 criteria on treatment. Per RECIST 1.1 for target lesions: CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. PR or better overall response assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and absence of new lesions.
Time Frame: Disease was evaluated radiologically at baseline, on trt every 6 weeks (wks) for the first 18 wks and then every 12 wks; Median (range) trt duration was 12 weeks (3-67).
Population: The analysis dataset is comprised of all treated patients.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Trastuzumab and Vinorelbine - Cohort A | Trastuzumab and Vinorelbine - Main Cohort
Number analyzed (Participants) | 11 | 20
percentage of patients | 18.2 [2.3 to 51.8] | 5.0 [0.1 to 24.9]

2. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: CBR was defined as achieving complete response (CR), partial response (PR), or stable disease (SD) for 24 weeks or longer based on RECIST 1.1 criteria on treatment. Per RECIST 1.1 for target lesions: CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. PD is at least a 20% increase in sum LD of target lesions (smallest sum LD reference), new lesions, and/or unequivocal progression of existing non-target lesions. Stable disease (SD) is defined as any condition not meeting the above criteria. SD needed to be a minimum 24 weeks in duration
Time Frame: as for outcome 1
Population: The analysis dataset is comprised of all treated patients.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Trastuzumab and Vinorelbine - Cohort A | Trastuzumab and Vinorelbine - Main Cohort
Number analyzed (Participants) | 11 | 20
percentage of patients | 63.6 [30.8 to 89.1] | 20.0 [5.7 to 43.7]

3. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS based on the Kaplan-Meier method is defined as the duration of time from study entry to documented disease progression (PD) requiring removal from the study or death. Per RECIST 1.1 for target lesions: PD is at least a 20% increase in sum LD, taking as reference the smallest sum on study with at least 5 mm absolute increase. For non-target lesions, progression-free means no new lesions or unequivocal progression on existing non-target lesions or not evaluated.
Time Frame: Disease was evaluated radiologically at baseline, on trt every 6 weeks (wks) for the first 18 wks and then every 12 wks and within 2 wks off-study; Median follow-up was 2.7 months.
Population: The analysis dataset is comprised of all treated patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab and Vinorelbine - Cohort A | Trastuzumab and Vinorelbine - Main Cohort
Number analyzed (Participants) | 11 | 20
months | 6.9 [5.4 to NA] — Follow-up is not long enough/Data is not mature to provide upper bound 95% confidence interval (CI). | 2.7 [2.6 to NA] — Follow-up is not long enough/Data is not mature to provide upper bound 95% CI.

4. Secondary Outcome: Baseline Level of Circulating Tumor Cells (CTCs)
Description: CTCs levels were determined based on established methods.
Time Frame: Assessed at baseline
Population: The CTCs in cohort A were analyzed using a non-CLIA approved assay and thus it was felt that the outcome data for this cohort were not evaluable. A new CLIA approved assay was used for the main cohort.
Measure: Median (Full Range); unit: cells per 7.5 ml blood
Arm/Group | Trastuzumab and Vinorelbine - Main Cohort
Number analyzed (Participants) | 20
cells per 7.5 ml blood | 5.5 [1 to 249]

ADVERSE EVENTS:
Time Frame: Assessed day 1 of each cycle throughout treatment. Median follow-up was 2.7 months.
Description: Based on common terminology criteria for adverse events version 4(CTCAEv4), maximum grade toxicity by type was first calculated for AEs with trastuzumab and/or vinorelbine treatment-attribution of possibly, probably or definite. Grade 3 or higher AEs were classified as serious and grade 1-2 AEs were classified as other. No further data is available to specify classification of other beyond the general term.
Arm/Group | Trastuzumab and Vinorelbine - Cohort A | Trastuzumab and Vinorelbine - Main Cohort
Serious Adverse Events (participants affected / at risk) | 9/11 | 11/20
Other Adverse Events (participants affected / at risk) | 11/11 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab and Vinorelbine - Cohort A (N=11) | Trastuzumab and Vinorelbine - Main Cohort (N=20)
Abdominal infection (Infections and infestations) | 0 | 1
Allergic reaction (Immune system disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 2 | 1
Ascites (Gastrointestinal disorders) | 1 | 0
Cardiac disorders - Other, specify (Cardiac disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Creatinine increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Fatigue (General disorders) | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Infections and infestations - Other (Infections and infestations) | 2 | 0
Intracranial hemorrhage (Nervous system disorders) | 1 | 0
Investigations - Other (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 1 | 0
Mediastinal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 1 | 0
Neutrophil count decreased (Investigations) | 7 | 4
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab and Vinorelbine - Cohort A (N=11) | Trastuzumab and Vinorelbine - Main Cohort (N=20)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 4
Alkaline phosphatase increased (Investigations) | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2
Anemia (Blood and lymphatic system disorders) | 6 | 8
Anorexia (Metabolism and nutrition disorders) | 0 | 5
Anxiety (Psychiatric disorders) | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 6
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Bloating (Gastrointestinal disorders) | 1 | 0
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0
Blurred vision (Eye disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Breast pain (Reproductive system and breast disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 2 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Creatinine increased (Investigations) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 3 | 0
Diarrhea (Gastrointestinal disorders) | 3 | 4
Dizziness (Nervous system disorders) | 2 | 1
Dry eye (Eye disorders) | 2 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2
Duodenal hemorrhage (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 3
Dysphagia (Gastrointestinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 8
Edema limbs (General disorders) | 2 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2 | 0
Fatigue (General disorders) | 8 | 13
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 2
Fecal incontinence (Gastrointestinal disorders) | 1 | 0
Fever (General disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Flatulence (Gastrointestinal disorders) | 1 | 0
Floaters (Eye disorders) | 0 | 1
Flu like symptoms (General disorders) | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 | 4
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 | 0
General disorders and administration site conditions - Other (General disorders) | 0 | 1
Headache (Nervous system disorders) | 3 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 0
Hepatobiliary disorders - Other (Hepatobiliary disorders) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 3
Hypertension (Vascular disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Infusion related reaction (General disorders) | 1 | 1
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 1 | 0
INR increased (Investigations) | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 2
Laryngitis (Infections and infestations) | 1 | 0
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 2 | 0
Mucositis oral (Gastrointestinal disorders) | 1 | 3
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 3 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 3 | 7
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Neutrophil count decreased (Investigations) | 1 | 4
Non-cardiac chest pain (General disorders) | 1 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Otitis media (Infections and infestations) | 1 | 0
Pain (General disorders) | 3 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Paronychia (Infections and infestations) | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 1 | 5
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 4
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 | 0
Sinusitis (Infections and infestations) | 1 | 0
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 | 1
Skin infection (Infections and infestations) | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Urinary urgency (Renal and urinary disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2
Weight loss (Investigations) | 0 | 2
White blood cell decreased (Investigations) | 1 | 1

LIMITATIONS AND CAVEATS:
The study terminated early due to insufficient response per statistical design.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No